CLINICAL TRIAL: NCT04073602
Title: An Open-label, Single-arm, Single-center, Phase II Study to Evaluate the Efficacy and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate for Injection in Subjects With HER2-negative Metastatic or Unresectable Urothelial Cancer
Brief Title: A Study of RC48-ADC in Subjects With HER2-negative Locally Advanced or Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C011
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): Participants will be treated with RC48-ADC 2.0 mg/kg, once every 2 weeks (Q2W) until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — The eligible patients will be treated with RC48-ADC, an antibody-drug conjugate, 2.0 mg/kg, once every two weeks until investigator-assessed loss of clinical benefit, unacceptable toxicity, investigator or participant's decision to withdraw from therapy, or death (whichever occurs first).
  Other Names: Recombinant Humanized anti-HER2 Monoclonal Antibody-MMAE Conjugate For Injection

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in patients with locally advanced or metastatic HER2-negative urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Diagnosed with histologically or cytologically-confirmed locally advanced or metastatic urothelial cancer, originate from bladder, renal pelvis, ureter and urinary tract.
* Unresectable or disease progression (i.e. locally advanced/metastasis) after surgery and at least regular chemotherapy including gemcitabine, cisplatin AND paclitaxel. Disease progression within 6 months of the completion of neo-adjuvant and adjuvant chemotherapy with gemcitabine, cisplatin AND paclitaxel is also eligible.
* Measurable lesion according to RECIST 1.1.
* HER2 negative (i.e. IHC -or 1+) as confirmed by the department of Pathology in Beijing Cancer Hospital. Subject is able to provide specimens from primary or metastatic lesions for HER2 tests.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment:

Cardiac ejection fraction ≥ 50 %. Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5×10^9/L Platelets ≥ 100×10^9/L; Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN and ≤ 5 x ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN.

* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Known hypersensitivity to the components of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate.
* Toxicity of previous anti-tumor treatment not recovered to CTCAE Grade 0-1 (with exception of Grade 2 alopecia).
* Pleural or abdominal effusion with clinical symptoms that requires ongoing treatment.
* History of receiving any anti-cancer drug/biologic treatment within 3 weeks prior to trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* Currently known active infection with HIV or tuberculosis.
* Diagnosed with HBsAg , HBcAb positive and HBV DNA copy positive, or HCVAb positive.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 3 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* known central nervous system metastases.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.
* NYHA Class III heart failure
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR)as assessed by Investigator | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  Tumor response was assessed by investigator according to RECIST v1.1
Duration of Objective Response (DOR) | 24 months
  DOR was defined as the time from first documented OR to first documented PD or death from any cause, whichever occurred earlier
Disease control rate (DCR) | 24 months
  DCR was defined as the proportion of patients who achieved an objective response or maintained stable disease during the study
Overall Survival(OS) | up to 24 months
  OS was defined as the time from the first study treatment to the date of death from any cause.
Adverse Events | 28 days after the last dose of study treatment
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan X, Li J, Xu H, Liu Y, Zhou L, Li S, Wu X, Tang B, Chi Z, Cui C, Si L, Mao L, Lian B, Wang X, Duan R, Li C, Fang J, Guo J, Sheng X. Efficacy and safety of DV in HER2-negative and HER2-low locally advanced or metastatic urothelial carcinoma: Results of a phase 2 study. Med. 2025 Jul 11;6(7):100637. doi: 10.1016/j.medj.2025.100637. Epub 2025 Mar 19. PMID 40112819